CLINICAL TRIAL: NCT03512457
Title: Effect of Skin Self-examination Education Delivered During the Mammography Experience.
Brief Title: Skin Self-Examination Education During Mammography
Acronym: SSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Sarah M. Friedewald, MD (Unknown); Jennifer N. Choi, MD (Unknown)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00207179
Record Dates: First submitted 2018-04-11; First posted 2018-04-30 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Melanoma
Keywords: Melanoma; Skin self-examination; mammogram
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Investigator
Masking Description: study arm not disclosed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Intervention (Experimental): Participants receive brochure, card advising how to make an appointment with dermatology, and reminder in one week to perform SSE.
  Interventions: Behavioral: Intensive Intervention
- Minimal Intervention (Active Comparator): Participants receive brochure, card advising how to make an appointment with dermatology, and reminder in one week to perform SSE.
  Interventions: Behavioral: Minimal Intervention

INTERVENTIONS:
Behavioral: Minimal Intervention — Women view an educational poster in changing room, and they receive a brochure.
  Arms: Minimal Intervention
Behavioral: Intensive Intervention — Women view an educational poster in changing room, and they receive a brochure.
  Arms: Intensive Intervention

SUMMARY:
The skin self-examination for melanoma (SSE) educational materials were developed with the input provided by women undergoing screening mammograms. The investigators seek to evaluate the performance of SSE by women and find out if women seek care with a dermatologist for a concerning mole or for a melanoma screening examination by a dermatologist after reviewing the materials received during the mammogram visit. The purpose of this study is to enhance the early detection of melanoma among women who are engaging in health promotion by having mammograms. The investigators specifically aim to evaluate the performance of SSE by women, who receive information during their mammogram appointment, and then follow-up with dermatology for a melanoma screening examination.

DETAILED DESCRIPTION:
The proposed study is the second phase of a project assessing the feasibility and effectiveness of enhancing the early detection of melanomas among women, who are engaging in health promotion by having mammograms. The initial phase of the project framed risk messages, developed posters and brochures with the input provided by women undergoing screening mammograms, and assessed the feasibility of delivering the program during the mammogram visit at the Lynn Sage Comprehensive Breast Center of Northwestern Medicine/ Prentice Women's Hospital. The investigators seek to evaluate performance of skin self-examination (SSE) by women, who receive information during their mammogram appointment, and follow-up with dermatology for a melanoma screening examination. In the second phase, a more intensive intervention in which women will not only receive information about SSE, but will also receive a reminder to perform SSE one week after the screening mammogram and information on how to schedule an appointment with dermatology will be provided. The number of women who perform SSE at home and find a concerning mole (lesion), number who see a dermatologist, and number who have a concerning lesion biopsied will be compared in two arms of the study 1) women who receive the intensive intervention 2) women who receive the informational brochure about SSE alone. The hypothesis is that women who receive more the intensive educational intervention will be more likely to perform SSE at home and schedule a follow-up dermatologist appointment as compared to those who receive the information brochure alone. This project builds upon Robinson's successful SSE training program for melanoma patients that resulted in patients' accurate evaluations of suspicious lesions relative to dermatologists' skin examinations.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Waiting to have a mammogram

Exclusion Criteria:

* Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women waiting to have a mammogram
Enrollment: 420 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: June K. Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rzepecki AK, Jain N, Ali Y, Chavez L, Choi J, Schlosser B, Liko-Hazizi E, Friedewald SM, Robinson JK. Promoting early detection of melanoma during the mammography experience. Int J Womens Dermatol. 2017 Jul 5;3(4):195-200. doi: 10.1016/j.ijwd.2017.06.002. eCollection 2017 Dec. PMID 29234713
- [Result] Robinson JK, Perez M, Abou-El-Seoud D, Kim K, Brown Z, Liko-Hazizi E, Friedewald SM, Kwasny M, Spring B. Targeted Melanoma Screening: Risk Self-Assessment and Skin Self-Examination Education Delivered During Mammography of Women. JNCI Cancer Spectr. 2019 Jun 28;3(3):pkz047. doi: 10.1093/jncics/pkz047. eCollection 2019 Sep. PMID 32328556
- [Derived] Robinson JK, Brown Z, Spring B. Melanoma Skin Self-Examination Education During Mammography: Health Burden of Women Impairs Implementation. J Cancer Educ. 2021 Aug;36(4):858-864. doi: 10.1007/s13187-020-01714-4. PMID 32090289

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Intervention: Participants receive brochure, card advising how to make an appointment with dermatology, and reminder by telephone, text message or email in one week to perform SSE.
  Intensive Intervention: Women view an educational poster in changing room, and they receive a brochure.
- Minimal Intervention: Participants receive brochure, card advising how to make an appointment with dermatology.
  Minimal Intervention: Women view an educational poster in changing room, and they receive a brochure.
Period: Overall Study
Arm/Group | Intensive Intervention | Minimal Intervention
Started | 195 | 225
Completed | 161 | 185
Not Completed | 34 | 40

BASELINE CHARACTERISTICS:
Population: Women having a screening mammogram completed a baseline self-report of prior skin self-examination prior to the intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Intervention | Minimal Intervention | Total
Number analyzed (Participants) | 195 | 225 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.9) | 53.1 (9.9) | 52.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 225 | 420
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 15 | 37
  Not Hispanic or Latino | 173 | 210 | 383
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 30 | 43 | 73
  White | 140 | 162 | 302
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 12 | 9 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 195 | 225 | 420
Number of participants who had ever conducted skin self-examination prior to study participation [Count of Participants; unit: Participants] | 55 | 70 | 125

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Performed a Skin Self-Examination at 3-months
Description: The percentage of participants that performed skin self-examination at the 3-month time interval.
Time Frame: 3-months
Population: Women performing skin self-examination as reported 3 months after the intervention
Measure: Count of Participants; unit: Participants
Groups:
- Intensive Intervention: Women who received an educational brochure and a 1-week reminder call or email to complete SSE
- Educational Intervention: Women who only received a brochure.
Arm/Group | Intensive Intervention | Educational Intervention
Number analyzed (Participants) | 195 | 225
Participants | 161 | 185
Statistical Analysis 1: Comparison: Intensive Intervention vs Educational Intervention; change from baseline to 3 months in performance of skin self-examination Parallel: response rate; Test type: Superiority — Chi-square; p = 0.12, Chi-squared — P-value of <0.05 is the threshold for statistical significance. The hypothesis was that more women randomized to the intensive intervention would perform skin self-examination; Chi-Squared is equal to 1.58, with a P-Value of 0.12

2. Secondary Outcome: Total Number of Melanomas Determined by Dermatologist Review of Concerning Lesion
Description: The total number of melanomas identified by a dermatologist in women who found a concerning mole
Time Frame: 7-months
Population: Women who found a concerning mole at month 1 and month 3 and proceeded to have a skin examination by a dermatologist
Measure: Number; unit: Melanomas
Arm/Group | Intensive Intervention | Minimal Intervention
Number analyzed (Participants) | 20 | 23
Melanomas | 2 | 5
Statistical Analysis 1: Comparison: Intensive Intervention vs Minimal Intervention; results of skin clinical examination and biopsy of clinically suspicious moles; Test type: Superiority — Types of lesions in the following categories: Benign nevus, seborrheic keratosis, lentigo, dermatofibroma, atypical nevus. melanoma; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 7 months
Groups:
- Intensive Intervention: Participants receive brochure, card advising how to make an appointment with dermatology, and reminder in one week by telephone call, text message or email to perform SSE.
  Intensive Intervention: Women view an educational poster in changing room, and they receive a brochure.
Arm/Group | Intensive Intervention | Minimal Intervention
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/225
Serious Adverse Events (participants affected / at risk) | 0/195 | 0/225
Other Adverse Events (participants affected / at risk) | 0/195 | 0/225

LIMITATIONS AND CAVEATS:
Limitations of our study include a relatively short duration of follow-up resulting in a modest number of incident invasive melanoma cases and a lack of participant blinding of allocation to intervention arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03512457/Prot_SAP_000.pdf